CLINICAL TRIAL: NCT06457321
Title: Implementation of Digital Workflow for Complete Dentures - A Crossover Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Dental Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 370-2022
Record Dates: First submitted 2024-04-04; First posted 2024-06-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: Complete Edentulism
Keywords: Complete edentulism; Complete denture; Digital Denture; Computer aided design; Computer aided manufacturing; CAD; CAM
MeSH Terms: interventions — Base Sequence

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 2 groups which receive dentures fabricated by two different methods.
  Group 1: Participants receive denture made from Conventional method, followed by denture made from partial digital method Group 2: Participants receive denture made from partial digital method, followed by denture made from conventional method
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Receive conventionally made denture first then denture made from partial digital method. (Other): Participants will be receiving their Denture 1 made from conventional method first and provide feedback at the 1-month and 2-month Denture 1 post-issue review visits.
  Participants will then return the Denture 1 to the attending clinician and receive the Denture 2 made from partial digital method and provide feedback at the 1-month and 2-month post-issue Denture 2 review visits.
  Interventions: Procedure: Sequence in receiving the fabricated dentures made using the conventional and partial digital method
- Receive denture made from partial digital method first then conventionally made denture. (Other): Participants will be receiving their Denture 1 made from partial digital method first and provide feedback at the 1-month and 2-month Denture 1 post-issue review visits.
  Participants will then return the Denture 1 to the attending clinician and receive the Denture 2 made from conventional method and provide feedback at the 1-month and 2-month post-issue Denture 2 review visits.
  Interventions: Procedure: Sequence in receiving the fabricated dentures made using the conventional and partial digital method

INTERVENTIONS:
Procedure: Sequence in receiving the fabricated dentures made using the conventional and partial digital method — Participants is not informed on the sequence they have been randomized hence they are not able to determine which denture is fabricated from which method. This would reduce bias when collecting the participants' responses in the satisfaction questionnaire during the review visits.

SUMMARY:
With a demographically ageing population and increasing patients with missing teeth, the demands on the healthcare system are set to further increase. This project is to prepare the public dental healthcare system to remain sustainable in terms of efficiency of denture production and healthcare manpower (lab technicians, clinician and operation staff). It aims to understand and improve denture fabrication productivity, enhance the treatment efficiency. This new model of care is a change from the current staged treatment process to batch processing assisted by new manufacturing methods, with the goal of improving sustainability and effectiveness of existing clinical and dental lab capacities.

DETAILED DESCRIPTION:
With an ageing population and growing demand for denture treatments, the conventional denture manufacturing method is incapable of meeting the current demand in Singapore due to its labour intensity and low efficiency. Such a growing demand urgently necessitates simplification and automation in denture manufacturing. Study team propose to deploy and pilot implement a computer-aided design and computer aided manufacturing approach to fabricate the complete dentures. With this innovative, automated manufacturing approach, study team will be able to produce the dentures in a couple of days, improve clinical efficiency, reduce lab production time and manpower needed. The digital workflow will be able to decrease the reliance on technical skills and thus reduce human variation and error and substantially enhance denture fabrication productivity. Successful implementation of this innovative denture manufacturing approach will lead to more timely and cost-effective access to denture care for many older Singaporeans, thus improving their quality of life.

This proposal aims to 1) to evaluate the cost and time used with both digital and conventional workflows; 2) to compare clinical outcomes between digital and conventional dentures; 3) to evaluate patients' satisfaction toward the digital dentures.

The long-term goal of this study is to reduce treatment cost and time, improve service efficiency and eventually enhance oral function and overall quality of life of complete edentulous patients.

Participants will be randomized into 2 groups to determine the sequence of the workflow:

Group 1: Conventional then partial digital Group 2: Partial digital than conventional

For conventional method

1.1 Clinical Examination

Informed consent will be obtained when patients attend the first visit for examination and diagnosis. Detailed examination of the oral mucosa and alveolar ridge will be carried out during the initial visit.

For conventional workflow, primary impressions using alginate impression material will be made with a stock tray for both maxillary and mandibular arches. This impression will be poured as a preliminary stone cast for fabrication of a PMMA resin custom impression tray in a conventional dental laboratory.

Participant will also be asked to complete questionnaires to rate their current denture:

During Fabrication (Visit 1-4)

* 3D Denture Patient Questionnaire OHIP EN (Pre-issue)
* 3D Denture Patient Questionnaire VAS

1.2 Master Impression

The customized special tray will be checked in patient mouth for fit and extension followed by border moulding using low fusing impression compound. Master impressions will be taken using special trays and zinc oxide impression paste or silicone materials. Stone casts will be created using green stone in the dental laboratory. The wax base will be constructed on the master models and wax rim will be added.

1.3 Jaw Relation Registration

Adjustment of wax rim will be made by clinicians to determine the vertical jaw relation, occlusal plane, and lip support. The size and shade of the teeth will be selected. The models will be mounted in the laboratory and teeth set up will be completed.

1.4 Aesthetic Try-in

The anterior and posterior teeth setup will be verified intraorally in patient. Maxillary and mandible relation will be confirmed. The articulator will be returned to the lab technician for finishing. The final dentures will be fabricated using the polymerizing polymethylmethacrylate resin, trimmed and polished by the dental technician.

1.5 Issue of denture

Necessary adjustments may be made by clinicians to meet the retention, stability and support requirements. The finished complete dentures will be evaluated in the patient mouth. Patients will be invited to fill in the questionnaire to report on oral health related quality of life (OHRQoL) and chewing ability based on the usage of patients' existing dentures.

1.6 Follow-up visits

Patients will be followed up two times at 2 weeks and 4 weeks after dentures are issued. Necessary modifications to the dentures will be made to ensure the comfort and function of the devices. Patients' oral health related quality of life and general satisfaction with the complete dentures, including aesthetics, retention, speech, chewing and comfort will be assessed using a self-administered questionnaire .

For partial digital method

2.1 [Clinic] Informed consent will be obtained when the patients attend their first visit for examination and diagnosis upon being called. Detailed examination of the oral mucosa and alveolar ridge will be carried out in the initial visit. Like the conventional workflow, primary impressions with an alginate impression material will be used with a stock tray for both maxillary and mandibular arches. This impression will be used to pour a preliminary stone cast.

[Lab] The preliminary stone cast will be thereafter scanned digitally using a lab scanner. Design of special tray will be carried out on the computer programme and 3D printing of PMMA resin custom impression tray will be conducted using a resin printer. A wax rim can then be conventionally added on top of this resin tray for the next visit.

2.2 Master Impression + Maxillomandibular Registration

[Clinic]The customized special tray will be checked in patient mouth for fit and extension followed by border moulding using low fusing impression compound. Master impressions will be taken using special trays and an addition polymerization silicone material. The OVD and maxillomandibular relationship will also be recorded using the wax rims and bite registration material during this visit.

[Lab] The master impression on the intaglio surface and registered wax rim will be scanned using an intra-oral scanner. Subsequently, the digital set-up of the denture teeth will be done. This preliminary teeth set up is then printed in resin for a try in during the next visit.

2.3. Aesthetic Try-in

[Clinic] The anterior and posterior teeth setup will be verified intraorally in patient. Maxillomandibular relationship and aesthetics relation will be verified. If changes are required, clinicians will be able to trim the resin teeth and base to achieve adequate maxillary and mandible relationship.

[Lab] The eventual verified MMR relationship will be scanned again. Adjustments to the digital teeth set up can be adjusted where necessary. The final dentures will be printed using the polymerizing polymethylmethacrylate resin, trimmed and polished by the dental technician.

2.4 Issue of denture

Necessary adjustments may be made by clinicians to meet the retention, stability and support requirements. The finished complete dentures will be evaluated in the patient mouth. Patients will be invited to fill in the questionnaire to report on oral health related quality of life (OHRQoL) and chewing ability based on the usage of patients' existing dentures.

2.5 Follow-up visits

Patients will be followed up two times at 2 weeks and 4 weeks after dentures are issued. Necessary modifications to the dentures will be made to ensure the comfort and function of the devices. Patients' oral health related quality of life and general satisfaction with the complete dentures, including aesthetics, retention, speech, chewing and comfort will be assessed using a self-administered questionnaire .

Sequence of issue

The patients will be randomised into 2 groups, determining the sequence in which the 2 sets of dentures from both workflows will be issued. The initial denture treatment stages from both workflows will be done concurrently. However, depending on which group they have been randomised into, they will be issued the conventional of the partial digital denture first.

After reviewing the patient thrice (at 2 weeks, 4 weeks and 2 months) for adjustments where necessary, the second set of denture from the other workflow will be issued and reviewed at the same time intervals. This allows ample time for the patient to test out and adapt to each set of denture from both workflows.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete edentulism requiring complete denture treatments.
* Prior denture experience.
* Above the age of 21 years.
* Medically fit (ASA classification of physical status I-III);
* Able to write/read English or Chinese well.

Exclusion Criteria:

* New denture wearers.
* Patients require surgical interventions to correct ridge anatomy.
* Patients with a history of maladaptation to denture use.
* Patients with maxillofacial defects.
* Patients unable to response to the English/Chinese questionnaires.
* Patients with enlarged tuberosity, minimal bone resorption resulting in limited restorative space
* Patients with enlarged tori
* Patients with flabby ridge
* Patients with severely resorbed ridges
* Patients with severe skeletal relationship discrepancy

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients' Oral Health Quality of Life | End of 2 months review of Denture 1 and Denture 2 respectively
  To investigate patients' perceived oral health related quality of life (OHRQoL) by comparing patients' responses after receiving complete dentures fabricated by conventional or digital workflows.
  This will be completed at 5 time points:
  1. before receiving Denture 1
  2. 4 weeks after using Denture 1
  3. 2 months after using Denture 1
  4. 4 weeks after using Denture 2
  5. 2 months after using Denture 2
  Denture 1 and 2 can be either conventionally made denture or denture made from partial digital method.
  There are a total of 14 questions and each question has 5 options to choose from and scores are tagged to the options ranging from 0 to 4. The total minimum and maximum score for each attempt is 0 and 56 respectively. The higher the score, the worser the QoL.
Patients' Denture Satisfaction | End of 2 months review of Denture 1 and Denture 2 respectively
  To investigate patients' satisfaction towards the denture fabricated using the McGill Denture satisfaction questionnaire by comparing patients' responses after receiving complete dentures fabricated by conventional or digital workflows.
  The set of questionnaires will have to be completed at 5 time points:
  1. before receiving Denture 1
  2. 4 weeks after using Denture 1
  3. 2 months after using Denture 1
  4. 4 weeks after using Denture 2
  5. 2 months after using Denture 2
  Denture 1 and 2 can be either conventionally made denture or denture made from partial digital method.
  There are a total of 26 questions and each question has a scale from 0 to 100. Participants can then give a score.
  0 - implies extremely not satisfied. 100 - implies extremely satisfied. The total minimum and maximum score for each attempt of this questionnaire is 0 and 2600 respectively. The higher the score, the higher the satisfaction from the patients on their denture.

SECONDARY OUTCOMES:
Cost saving | From start of fabrication to the issue of the denture to participants, up to 8 months
  To calculate the cost saved by the number of visits that the patients have to fulfill and also the material cost to see if one is significantly more affordable than the other.
Time efficiency | From start of fabrication to the issue of the denture to participants, up to 8 months
  To measure the time taken to fabricate the dentures using the two methods to see if one is significantly shorter than the other.

IPD SHARING:
Plan to Share IPD: No